CLINICAL TRIAL: NCT01044875
Title: A Randomised Control Trial Comparing the Effectiveness of Yellow 577 nm Laser to Conventional Green 532 nm Laser for Proliferative Diabetic Retinopathy
Brief Title: Trial of Yellow 577 nm Laser Versus Green 532 nm Laser for Proliferative Diabetic Retinopathy
Acronym: UMPDR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Malaya (Other)
Responsible Party: Assoc Prof Kenneth C S Fong, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UMERC002
Record Dates: First submitted 2010-01-07; First posted 2010-01-08 (Estimated); Last update posted 2010-01-08 (Estimated); Status verified 2010-01

CONDITIONS: Proliferative Diabetic Retinopathy
Keywords: Diabetic retinopathy; Laser treatment; Complications; Laser wavelength
MeSH Terms: conditions — Diabetic Retinopathy | interventions — Lasers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- green laser 532 nm conventional (Active Comparator): Current type of laser used for treatment of proliferative diabetic retinopathy
  Interventions: Procedure: Pan retinal photocoagulation laser treatment
- Yellow 577 nm laser (Active Comparator): new laser wavelength for treatment of PDR
  Interventions: Procedure: Pan retinal photocoagulation laser treatment

INTERVENTIONS:
Procedure: Pan retinal photocoagulation laser treatment — Eyes with PDR are randomised to treatment with either the green laser 532 nm or 577 nm yellow laser.
  Other Names: Quantel Supra 577nm laser

SUMMARY:
The purpose of this study is to measure effectiveness of yellow 577 nm laser compared to conventional green laser 532 nm for diabetic retinopathy in terms of number of treatment sessions required and visual acuity outcome.

The study also compares pain score of patients receiving laser treatment and side effects of laser treatment.

DETAILED DESCRIPTION:
Diabetes mellitus (DM) is a major medical problem throughout the world. The most common and potentially most blinding of these complications is proliferative diabetic retinopathy (PDR).

Panretinal photocoagulation is established as the gold standard of treatment, supported by the data of the Diabetic Retinopathy Study (DRS).This study found that laser treatment reduced the rate of severe visual loss by 50%. Currently the green 532nm laser is the most common wavelength used. However, this conventional green laser has some complications such as pain, vitreous haemorrhage, choroidal effusion and visual field loss.

Due to the complication of conventional lasers, the yellow laser (577 nm)with peak absorption of oxyhemoglobin and good absorption of melanin is postulated to be more effective at producing retinal laser burns with a lower power and less pain compared to the green laser.

ELIGIBILITY:
Inclusion Criteria:

* Patient more than 18 year of age
* Eyes with proliferative diabetic retinopathy requiring laser PRP
* Newly diagnosed patient
* Patients with no other intervention/surgeries done before the study

Exclusion Criteria:

* Eyes with media opacity not allowing adequate laser photocoagulation
* Patients who have had previous laser photocoagulation
* Patients who have had previous vitreoretinal surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2009-09; Primary Completion 2011-09 (Estimated); Study Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
Visual acuity measurement by logarithm of the minimum angle of resolution (logMAR) | 2 years

SECONDARY OUTCOMES:
Patient pain score during laser procedure | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth C Fong, FRCOphth, Principal Investigator — University of Malaya Eye Research Centre; Nurliza Khaliddin, FRCS, Principal Investigator — University of Malaya Eye Research Centre
Locations (1):
- University of Malaya Eye Research Centre, Kuala Lumpur, Kuala Lumpur, Malaysia